CLINICAL TRIAL: NCT01706731
Title: A Randomized Controlled Trial of Cognitive Behavior Therapy Provided by Buddhist Monks vs. Treatment as Usual in the Treatment of Late Life-depression
Brief Title: Effectiveness of Buddhist Monks in Providing Cognitive Behavior Therapy
Acronym: Add-CBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Nahathai Wongpakaran, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 918
Record Dates: First submitted 2012-10-08; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Major Depressive Disorder
Keywords: Buddhist monks; CBT; elderly; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU plus Cognitive-behavioral Therapy (Active Comparator): Participants randomized to this group will receive treatment as usual plus cognitive behavioral therapy (CBT) provided by trained Buddhist monks.
  Interventions: Behavioral: Treatment as usual; Behavioral: Cognitive-behavioral therapy
- TAU plus routine counselling (Sham Comparator): Participants randomized into this group will receive treatment as usual (TAU) plus plus routine psychological support from non-CBT monks.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Treatment as usual — Treatment as usual (TAU)is defined as the routine care provided to each individual patient at the geriatric psychiatry clinic of Maharaj Nakorn Chiang Mai Hospital.
  Other Names: TAU
Behavioral: Cognitive-behavioral therapy — Cognitive behavioral therapy(CBT)includes psychoeducational components combined with cognitive interventions targeted at challenging negative automatic thoughts.
  Arms: TAU plus Cognitive-behavioral Therapy

SUMMARY:
This research is to study the effectiveness of cognitive behavioral therapy-CBT and Psychotherapy by trained buddhist monks. There are generally accepted that both cognitive and Buddhist concepts are related. This randomized controlled trial is to study the elderly participants who suffer major depressive disorder according to DSM-IV. The subjects will be divided into two groups. The experimental group will receive 12 sessions of CBT 2 times per week for 6 weeks in addition to usual treatment. The control group will receive treatment as usual and general conversation (non-CBT) with monks. Pretreatment factors (such as attachment style, interpersonal factors) of both therapist monks and patient participants will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for Major depressive disorder
* receiving antidepressant

Exclusion Criteria:

* presence of intense suicidal intent behaviors that require inpatient admission
* history of alcohol or drug dependence
* presence of hallucinations or delusions
* currently receiving electroconvulsive therapy or repetitive-transcranial magnetic stimulation,
* patients' involvement in other clinical trials.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically depression confirmed by clinician | 2 months after the end of the intervention
  Depression will be assessed by HAMD-7 (McIntyre, 2005)
Depression- self report | 2 month after the end of the inetrvention
  depression will be assessed by Geriatric Depression Scale (GDS)(Shiekh & Yesavage, 1986)

SECONDARY OUTCOMES:
Dimensional psychological distress (anxiety, depression,and somatization) | week 6, 12, 20
  anxiety, depression,and somatization symptom will be assessed by the Core symptom index (CSI) (Wongpakaran, unpublished),
Dimensional psychological distress ( perception of stress) | Week 6, 12, 20
  Perception of stress will be assessed by Perceived Stress Scale-10 (PSS-10) (Cohen 1983 ; Wongpakaran, 2010)

OTHER OUTCOMES:
working alliance | after session 3, 6, and 12
  Working alliance will be assessed by the Helping Alliance Questionnaire (HAQ)(Luborsky, 1996)
Pretreatment measure (attachment) | at baseline
  The part includes participants' attachment which will be assessed by the revised Experience of Close Relationships Questionnaire (ECR-R 18)(Wongpakaran, 2012)
Pretreatment measure (interpersonal problems) | at baseline
  Interpersonal problems will be assessed by the inventory of interpersonal problems(Horowitz, 2000)
Pretreatment measure(neuroticism) | at baseline
  Neuroticism will be assessed by the Neuroticsm Inventory (Wongpakaran,unpublished)

CONTACTS AND LOCATIONS:
Overall Officials: Nahathai - Wongpakaran, M.D., Principal Investigator — Chiang Mai University
Locations (1):
- Geriatric clinic, Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Chiang Mai, Thailand